CLINICAL TRIAL: NCT01062360
Title: A Pivotal, Placebo Controlled, Phase III Study to Compare Efficacy and Tolerability of a Fixed Combination, Containing 500 mg ASA and 30 mg Pseudoephedrine, in Comparison to Its Single Components in Patients With Sore Throat and Nasal Congestion
Brief Title: Placebo and Active Controlled Study to Assess Efficacy and Tolerability of Aspirin Plus Pseudoephedrine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11764; 2005-001720-36 (EudraCT Number)
Record Dates: First submitted 2009-12-09; First posted 2010-02-04 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Common Cold; Pharyngitis
Keywords: Sore Throat; Upper Respiratory Tract Infections; Nasal Congestion
MeSH Terms: conditions — Common Cold; Pharyngitis; Respiratory Tract Infections; Nasal Obstruction | interventions — Aspirin; Pseudoephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin Complex, BAYE4465) + Pseudoephedrine
- Arm 2 (Active Comparator)
  Interventions: Drug: Acetylsalicylic Acid (Aspirin, BAYE4465)
- Arm 3 (Active Comparator)
  Interventions: Drug: Pseudoephedrine
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Acetylsalicylic Acid (Aspirin Complex, BAYE4465) + Pseudoephedrine — Single oral dose of 1 to 2 Aspirin Complex sachets, each containing granules of 500 mg Acetylsalicylic Acid (ASA) and 30 mg Pseudoephedrine (PSE), to be taken orally after dissolving in a glass of water; to be repeated as needed every 6 hours for a period of not more than 3 days.
  Arms: Arm 1
Drug: Acetylsalicylic Acid (Aspirin, BAYE4465) — Single oral dose of 1 to 2 sachets Acetylsalicylic Acid, each containing granules of 500 mg Acetylsalicylic Acid (ASA), to be taken orally after dissolving in a glass of water; to be repeated as needed every 6 hours for a period of not more than 3 days.
  Arms: Arm 2
Drug: Pseudoephedrine — Single oral dose of 1 to 2 sachets Pseudoephedrine, each containing granules 30 mg Pseudoephedrine, to be taken orally after dissolving in a glass of water; to be repeated as needed every 6 hours for a period of not more than 3 days.
  Arms: Arm 3
Drug: Placebo — Single oral dose of 1 to 2 sachets, each containing Placebo granules, to be taken orally after dissolving in a glass of water; to be repeated as needed every 6 hours for a period of not more than 3 days.
  Arms: Arm 4

SUMMARY:
The purpose of this study is compare efficacy and tolerability of a fixed combination, containing 500 mg Acetylsalicylic acid and 30 mg Pseudoephedrine, in comparison to its single components in patients with sore throat and nasal congestion.

ELIGIBILITY:
Inclusion Criteria:- Male and female subjects between 18 and 65 years of age.- Onset of cold symptoms within 96 hours (4 days) before study participation.- Current complaint of at least moderate sore throat at baseline- Current complaint of at least moderate NC at baseline- History of other symptoms associated with URTI during the last 4 days before study participation.- Other findings of URTI, confirmed on the physical examination.- Agreement to comply with the study requirements.- Written informed consent prior to enrollment in the study Exclusion Criteria:- Pregnant or lactating females.- Uncontrolled chronic diseases.- History of hypersensitivity (allergic reaction) to ASA, any other nonsteroidal anti-inflammatory drugs (NSAIDs), or PSE.- Any disease which significantly compromises breathing or interferes with the subjects assessment of sore throat.- History of or active peptic ulcer.- Severe impaired hepatic function.- Severe impaired renal function.- Simultaneous intake of monoamine oxidase inhibitors.- Use of menthol containing tissues within 2 hours before first intake of study drug.- Intake of any menthol containing product within 4 hours before first intake of study drug.- Use of any local or systemic short acting cough and cold preparations within 6 hours before first intake of study drug.- Use of any local or systemic long acting cough and cold preparations within 12 hours before first intake of study drug.- Intake of any analgesic within 12 hours before first intake of study drug.- Intake or requirement of any prescription medication for the treatment of the current acute respiratory tract infection.- Current or previous intake of anticoagulants, corticoids, NSAIDs, methotrexate, or lithium.- Participation in another clinical trial within the last 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1016 (Actual)
Dates: Start 2005-12-23 (Actual); Primary Completion 2007-05-14 (Actual); Study Completion 2007-05-14 (Actual)

PRIMARY OUTCOMES:
The primary efficacy parameter for the nasal congestion was the AUC calculated for baseline adjusted NCS for the initial 2 hours post dosing | 2 hours
The primary efficacy parameter for sore throat was SPID2 hours | 2 hours

SECONDARY OUTCOMES:
The Pain Intensity Difference at time point: 15, 30, 60, 90, 120, 240, and 360 minutes after the first dose | 15, 30, 60, 90, 120, 240, and 360 minutes
The Nasal Congestion Score | 15, 30, 60, 90, 120, 240, and 360 minutes
The Nasal Congestion Relief Score | 15, 30, 60, 90, 120, 240, and 360 minutes
Sore throat pain relief | 15, 30, 60, 90, 120, 240, and 360 minutes
The symptoms of common cold (headache, sinus pressure/pain, feverish discomfort, muscle aches, and pain) at 120 minutes post dose | 120 minutes
The results of an overall assessment of treatment by the subjects at 120 minutes post dose | 120 minutes
The results of an overall assessment of treatment by the subjects at the end of Day 3 after the first dose, or at the end of treatment (6 hours after last dose of study drug) | Day 3
Nasal Congestion, Pain Intensity Difference and pain relief at the end of Day 2 and at the end of Day 3, or at the end of treatment (6 hours after the last study drug intake) | Day 3
The symptoms of common cold (headache, sinus pressure/pain, feverish discomfort, muscle aches, and pain) at the end of Day 2 and at the end of Day 3, or at the end of treatment (6 hours after the last study drug intake) | Day 2 and Day 3
Total amount of drug intake | Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (35):
- New York, New York, United States
- Italy (20):
  - Alassio
  - Albenga
  - Arenzano
  - Civitella Marittima
  - Follonica
  - Genova
  - Grosseto
  - Grossetto
  - Isola del Cantone
  - Loano
  - Masone
  - Orbetello
  - Pegli
  - Quiliano
  - Rivarolo
  - Ronco Scrivia
  - Sampierdarena
  - Scansano
  - Serra Riccò
  - Varazze
- Poland (11):
  - Ciechocin
  - Dębowa Góra
  - Katowice
  - Krakow
  - Lodz
  - Piaseczno
  - Skierniewice
  - Szczecin
  - Torun
  - Warsaw
  - Zabrze
- Slovakia (3):
  - Bratislava
  - Pezinok
  - Stupava

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/